CLINICAL TRIAL: NCT04408378
Title: Retrospective Change in the Ratio of Mean Platelet Volume (MPV) to Platellet(PLT) in Covid-19 Pneumonia Patients
Brief Title: Change in the Ratio of Mean Platelet Volume (MPV) to Platellet(PLT) in Covid-19 Pneumonia Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gaziosmanpasa Research and Education Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: 69
Record Dates: First submitted 2020-05-27; First posted 2020-05-29 (Actual); Last update posted 2020-05-29 (Actual); Status verified 2020-05

CONDITIONS: Coronavirus Infection
Keywords: covid-19, MPV/PLT, pneumonia
MeSH Terms: conditions — Coronavirus Infections; COVID-19; Pneumonia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- mild pneumonia: The patients who has followed in the ward
  Interventions: Other: observation of covid 19 pneumonia
- severe pneumonia: The patiens who has followed in the intensive care unit
  Interventions: Other: observation of covid 19 pneumonia
- control group: patients who has not covid 19 pneumonia
  Interventions: Other: observation of covid 19 pneumonia

INTERVENTIONS:
Other: observation of covid 19 pneumonia — We try to reveal the fact,covid-19 pneumonia prognosis can be estimated by using MPV/PLT ratio

SUMMARY:
Morbidity, mortality and progress depends on systemic inflammation especially in ARDS patients. Previous studies claims that the proportion of mean platellet volume to platellet which can simply be determined with simple blood tests that are performed at admission, might predict the mortality in ARDS patients. Covid-19 pneumonia has a very similar clinical outlook with ARDS. Therefore we decided to research whether that proportion is legitimate for detecting the progress of Covid-19 pneumonia or not.

DETAILED DESCRIPTION:
Covid-19 pneumonia is a spesific disease dispate its similarity to ARDS. There are nomorous of studies that MPV/PLT ratio can predict the mortality, morbidity and the progress of ARDS. Depending on the similarity of ARDS, MPV/PLT ratio might predict the clinical progress of Covid-19 pneumonia. We retrospectively recruited150 patients admitted to our institute -a tertiary center- with Covid-19 pneumonia to our study. Clinical based defining research, by March-May 2020, the patients over 18 years old who were in either intensive care or ward scanned retrospectively. The laboratory tests, chronic diseases , age and gender has been collected from the written resources and electronic data retrospectively.

the patients who are diagnosed with Covid*19 pneumonia will be divided into two groups. The ones in the ward will be considered as mild clinical course, and the ones in the intensive care unit will be considered as severe clinical course. there will be an additional non Covid individuals as a control group, which will consist 52 patients each. The ratio of MPV to PLT will be calculated using admission hemogrames of these groups, and the significance of the statistical differences on determining the prognosis of the disease will be discussed.

Gpower 3 for Mac Os (Faul, F., Erdfelder, E., Buchner, A., & Lang, A.-G. (2009). Statistical power analyses using G*Power 3.1: Tests for correlation and regression analyses. Behavior Research Methods, 41, 11491160.) was used for istatistical power analysis.It was done using ANOVA test between at least two independent groups. In order to provide enoughsample magnitude power, which is 0.8, it was calculated that each group should have 52 patients which makes at total of 156.

The normal distribution of data will be evaluated using Kolmogorov-Smirnov test. Parametric ones will be used in normal distrubitions, non-parametric ones will be uused in abnormal distrubitions. Between the independent groups, MPV/PLT ratio will be calculated using ANOVA test. Categoric data will be compared by Pearson ki square test and the p values less than 0.05 will be considered as significant.

we aim to have an opinion about Covid 19-pneomonia prognosis at the admission of hospital.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old who hospitalized with diagnosis of Covid-19 pneumonia between march and may 2020

Exclusion Criteria:

* Under 18 years old patients
* Patients with heamolytic diaseses

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients over 18 years old who hospitalized with diagnosis of Covid-19 pneumonia between march and may 2020 in the ICU or ward.
Sampling Method: Probability Sample
Enrollment: 156 (Estimated)
Dates: Start 2020-06-05 (Estimated); Primary Completion 2020-07-20 (Estimated); Study Completion 2020-08-20 (Estimated)

PRIMARY OUTCOMES:
estimation of inflammatory changes in Covid 19 pneumonia by using MVP/PLT ratio | March-May 2020
  İt has been studied that MPV/PLT ratio can show the cl inical couses of several diseases as well as ARDS. we thought that we can identify the coronavirus pneumonia patients earlier, at admission of hospital by using the hemogrames.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaziosmanpaşa TREH, Istanbul, Gaziosmanpaşa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim CH, Kim SJ, Lee MJ, Kwon YE, Kim YL, Park KS, Ryu HJ, Park JT, Han SH, Yoo TH, Kang SW, Oh HJ. An increase in mean platelet volume from baseline is associated with mortality in patients with severe sepsis or septic shock. PLoS One. 2015 Mar 5;10(3):e0119437. doi: 10.1371/journal.pone.0119437. eCollection 2015. PMID 25742300
- [Background] Fei Y, Zhang H, Zhang C. The application of lymphocyte*platelet and mean platelet volume/platelet ratio in influenza A infection in children. J Clin Lab Anal. 2019 Nov;33(9):e22995. doi: 10.1002/jcla.22995. Epub 2019 Aug 16. PMID 31420904
- [Background] Korniluk A, Koper-Lenkiewicz OM, Kaminska J, Kemona H, Dymicka-Piekarska V. Mean Platelet Volume (MPV): New Perspectives for an Old Marker in the Course and Prognosis of Inflammatory Conditions. Mediators Inflamm. 2019 Apr 17;2019:9213074. doi: 10.1155/2019/9213074. eCollection 2019. PMID 31148950